CLINICAL TRIAL: NCT05615558
Title: The Impact of a High-Protein Diet From Animal vs. Non-Animal Sources on Insulin Sensitivity and β-cell Function in Type 2 Diabetes
Brief Title: High-Protein Diets and Diabetes
Acronym: HPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Collaborators: Marlow Foods Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 275134
Record Dates: First submitted 2022-05-26; First posted 2022-11-14 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Animal (Experimental): Arm of the study consuming a high-protein diet from animal sources.
  Interventions: Other: Dietary Intervention
- Non-animal (Experimental): Arm of the study consuming a high-protein diet from non-animal sources.
  Interventions: Other: Dietary Intervention

INTERVENTIONS:
Other: Dietary Intervention — Controlled dietary intervention; all food is provided to participants after being allocated to animal or non-animal dietary protein, for a duration of 5 weeks.

SUMMARY:
High-protein (HP) diets are popular and evidence indicates they are more likely to be adhered to and produce more sustained weight loss, particularly under ad libitum conditions. They also improve glucose control and so may be helpful for treatment of Type 2 Diabetes (T2D), particularly in the short-term, possibly via an improvement in insulin secretion. Indeed, HP diets may be uniquely effective at promoting insulin secretion in T2D, but further research is needed to understand why HP. Thus, there is an urgent need to determine how HP diets affect T2D pathophysiology of insulin secretion and action using direct measures of β-cell dysfunction and insulin sensitivity. It is also imperative to know how the type of protein (animal vs. non-animal) affects insulin secretion in order to ultimately obtain an environmentally and economically sustainable HP diet that can improve glucose control and T2D pathophysiology in the long-term as well as providing patients with a greater choice for dietary management of T2D.

ELIGIBILITY:
Inclusion Criteria:

* Aged 40-70 y
* Body-mass index of 27-45 kg/m2
* Diagnosed with T2D with their most recent HbA1c value greater than 6.0% (>43 mmol/mol) and receiving dietary advice and/or antidiabetic medication (metformin, DPP-4 inhibitors only).
* Males and females

Exclusion Criteria:

* Habitual dietary intake of <0.6 or >1.2 g/kg/day protein (determined from dietary history interview given at screening)
* Current use of insulin
* HbA1c of 12% or more (≥108 mmol/mol)
* Weight loss of more than 5 kg within the past 6 months
* A recent estimated glomerular filtration rate (eGFR) of less than 30 mL/min,
* Heart failure,
* Participation in another clinical research trial, substance abuse, known cancer, myocardial infarction within the previous 6 months, current treatment with anti-obesity drugs, pregnancy or consideration of pregnancy, and hospital admission for depression or use of antipsychotic drugs.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | Change from Baseline insulin sensitivity after 5-week controlled diet
  Rate of disappearance (Rd) during the hyperinsulinaemic-euglycaemic clamp from participants on each diet, a measure of insulin sensitivity.

SECONDARY OUTCOMES:
β-cell function | Change from Baseline β-cell function after 5-week controlled diet
  β-cell function measured by modelling of glucose, insulin and c-peptide during MMTT
Glucose control | Change from Baseline glucose control after 5-week controlled diet
  Glucose control measured by fasting glucose, 2 hour MMTT glucose, 24-hour glucose profile using continuous glucose monitoring probe and HbA1c.
Branched-chain amino acid (BCAA) metabolism | Change from Baseline BCAA after 1, 2, 3, 4 and 5 weeks of controlled diet
  BCAA metabolism measured by plasma BCAA concentration.
Diabetes treatment satisfaction measured by the diabetes treatment satisfaction questionnaire | Change from Baseline treatment satisfaction after 5-week controlled diet
  Treatment satisfaction measured by the diabetes treatment satisfaction questionnaire (DTSQ).

CONTACTS AND LOCATIONS:
Locations (1):
- Nutritional Physiology Research Unit, Exeter, Devon, United Kingdom